CLINICAL TRIAL: NCT01988883
Title: Modafinil and Cognitive Function in Postural Tachycardia Syndrome
Brief Title: Modafinil and Cognitive Function in POTS
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 131371; 5UL1TR000445-07 (NIH)
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Postural Tachycardia Syndrome
Keywords: Postural Tachycardia Syndrome; Tachycardia; Orthostatic Intolerance; Autonomic Nervous System Diseases; Primary Dysautonomias; Nervous System Diseases; Cardiovascular Diseases; Modafinil; Propranolol; Neurobehavioral Manifestations; Neurologic Manifestations; Cognitive Symptoms; Neuropsychological Tests
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Tachycardia; Orthostatic Intolerance; Autonomic Nervous System Diseases; Primary Dysautonomias; Nervous System Diseases; Cardiovascular Diseases; Neurobehavioral Manifestations; Neurologic Manifestations | interventions — Modafinil; Propranolol; propranolol CR

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Patients will receive two inactive placebo pills filled with microcrystalline cellulose on a randomized study day. Medications will be dummy blinded to the patient and investigators.
  Interventions: Drug: Placebo
- Modafinil (Experimental): Patients will receive single doses of modafinil (200 mg, oral) and placebo on a randomized study day. Medications will be dummy blinded to the patient and investigators.
  Interventions: Drug: Placebo; Drug: Modafinil
- Propranolol (Experimental): Patients will receive single doses of propranolol (20 mg, oral) and placebo on a randomized study day. Medications will be dummy blinded to the patient and investigators.
  Interventions: Drug: Placebo; Drug: Propranolol
- Modafinil plus Propranolol (Experimental): Patients will receive single doses of modafinil (200 mg, oral) and propranolol (20 mg, oral) on a randomized study day. Medications will be dummy blinded to the patient and investigators.
  Interventions: Drug: Modafinil; Drug: Propranolol

INTERVENTIONS:
Drug: Placebo — Locking gelatin capsules filled with microcrystalline cellulose
  Arms: Modafinil; Placebo; Propranolol
Drug: Modafinil — Modafinil is a wakefulness-promoting or psychostimulant drug. It will be administered as a single 200 mg oral tablet.
  Other Names: Provigil
  Arms: Modafinil; Modafinil plus Propranolol
Drug: Propranolol — Propranolol is a non-selective beta adrenergic antagonist.It will be administered as a single 20 mg oral tablet.
  Other Names: Inderal; Inderal LA; Innopran XL
  Arms: Modafinil plus Propranolol; Propranolol

SUMMARY:
A common complaint among patients with Postural Tachycardia Syndrome (POTS) is "brain fog" or difficulty concentrating. This problem is poorly understood.

The purpose of this study is to better understand the cognitive dysfunction associated POTS, and to determine optimal treatment strategies for this condition. In this study, the investigators will test the hypothesis that acute administration of the psychostimulant drug modafinil can improve seated measures of cognitive function in patients with POTS.

DETAILED DESCRIPTION:
Postural Tachycardia Syndrome (POTS) is one of the most frequent forms of chronic orthostatic intolerance and affects an estimated 500,000 people in the United States alone. This disorder is a common source of disability in young adults, with a strong predilection for premenopausal women. POTS is characterized by an excessive increase in heart rate (>30 bpm) on assuming the upright position that is associated with orthostatic symptoms that are relieved by lying down. These symptoms include palpitations, chest pain, lightheadedness or dizziness, blurred vision, nausea and fatigue. In addition, POTS patients commonly report mental clouding or "brain fog" even while lying down or seated, which can pose significant limitations to daily life.

Although mental clouding is an almost universal complaint among POTS patients, this phenomenon is poorly understood. As a result, the optimal treatment strategies to manage cognitive dysfunction in this condition remain unknown. The purpose of this study is to better define the mental clouding associated with POTS and to determine whether the psychostimulant modafinil is a viable therapeutic option to improve cognitive function in these patients. The investigators hypothesize that acute modafinil administration will improve seated measures of cognitive function in POTS patients. The specific aims are:

1. To assess whether acute modafinil improves seated measures of cognitive function, particularly measures of attention and executive function, in POTS patients compared to placebo.
2. To assess whether propranolol, either alone as an active control or in combination with modafinil to mitigate potential heart rate increases, can improve cognitive function in POTS.

Patients will be studied on 4 separate days with oral administration of: placebo, modafinil (200 mg), propranolol (20 mg) and the combination of modafinil (200 mg) and propranolol (20 mg). The order of administration will be randomized in a double-blind manner. Patients will be seated during the study and cognitive testing will begin approximately 2.5 hours after medication administration. Cognitive testing will consist of the CogState computerized brief battery. Patients will also be asked to stand for 10 minutes (or as long as tolerated) at 1, 3 and 4 hours post medication, with some of the cognitive tests repeated while standing at the 4 hour time point.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races between the ages of 18 to 60 years
* Diagnosed with POTS by the Vanderbilt Autonomic Dysfunction Center based on the following consensus criteria:(a) an increase in heart rate ≥ 30 beats per minute within 10 minutes of changing from the supine to standing position; (b) absence of orthostatic hypotension (defined as a decrease in systolic blood pressure ≥ 20 mmHg or diastolic blood pressure ≥ 10 mmHg upon standing); and (c) chronic symptoms (≥ 6 months) consistent with POTS that are worse with standing and are relieved by lying down
* Able and willing to provide informed consent

Exclusion Criteria:

* Overt causes for POTS such as acute dehydration and bed rest deconditioning
* Patients taking serotonin-norepinephrine reuptake inhibitors (SNRIs) or norepinephrine transporter (NET) inhibitors
* Known allergies or contraindications to study medications
* Pregnancy or breast-feeding
* Inability to give or withdraw informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the study protocol such as poor compliance during previous studies
* Asthma (due to the contraindication of propranolol for asthma patients)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Visual Attention Performance Speed | 2.5 hours post study medication
  This outcome will be assessed using the CogState Identification Task which provides a continuous variable for visual attention performance speed.

SECONDARY OUTCOMES:
Executive Function | 2.5 hours post study medication
  This outcome will be assessed by the CogState Groton Maze Learning and Set-Shifting Tasks which provides continuous variables for speed and accuracy measures of executive function.
Blood Pressure | Baseline and up to 4 hours after drug administration
  This outcome will be assessed using an automated sphygmomanometer arm cuff.
Heart Rate | Baseline and up to 4 hours after drug administration
  This outcome will be assessed using an automated sphygmomanometer arm cuff.

OTHER OUTCOMES:
Processing speed | 2.5 hours post study medication
  This outcome will be assessed by the CogState Detection task which provides continuous variables for speed and accuracy measures of processing speed.
Visual learning and memory | 2.5 hours post study medication
  This outcome will be assessed by the CogState One Card Learning task which provides continuous variables for speed and accuracy measures of visual learning and memory.
Working memory | 2.5 hours post study medication
  This outcome will be assessed by the CogState One-Back task which provides continuous variables for speed and accuracy measures of working memory.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States